CLINICAL TRIAL: NCT02590705
Title: Anesthesia Lumbar Puncture In Children (ALPIC)
Brief Title: Anesthesia Lumbar Puncture In Children
Acronym: ALPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Gang Liu, Chief physician/Professor, Beijing Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20150825
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Puncture; Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): surface anesthesia with lidocaine
  Interventions: Drug: Lidocaine
- Group 2 (No Intervention): no anesthesia

INTERVENTIONS:
Drug: Lidocaine — surface anesthesia with lidocaine
  Arms: Group 1

SUMMARY:
The study is carried out in a prospectively randomly controlled way. In the context of acknowledgement and understanding from parents, by comparing with traditional process(no anesthesia), lidocaine surface anesthesia is randomly selected. All children will be evaluated by the FLACC (The face, legs, activity, cry, consolability behavioral tool) scale to quantitatively assess degree of pain during lumbar puncture. Time and success rate of the lumber puncture will be recorded and analyzed. A questionnaire about bad memory during lumbar puncture for all parents and children will be investigated in order to establish an optimized lumbar puncture management process.

DETAILED DESCRIPTION:
The purpose of this study is to establish an optimized lumbar puncture management process on the basis of fully understanding of parents and children. An improved process consisting of painless lumbar puncture (LP) and comfortable LP will be established upon completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* children with indications of lumbar puncture;
* voluntarily signed the informed consent

Exclusion Criteria:

* topical anesthetic skin allergies;
* skin infection in lumbar puncture site;
* severe intracranial hypertension;
* unstable vital signs;
* coagulopathy;
* intracranial hemorrhage and occupying;
* low back pain;
* headache and low back pain before lumbar puncture;
* past headache after lumbar puncture;
* mental retardation, neuropsychiatric symptoms;
* children could not immediately act after the lumbar puncture(such as disturbance of consciousness or suffering from underlying diseases or drainage);
* the case with repeated puncture in one operation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
degree of adaptability | intraoperative
  evaluated by the FLACC(The face,legs,activity,cry,consolability behavioral tool) scale

SECONDARY OUTCOMES:
time of lumbar puncture | intraoperative
number of puncture | intraoperative
success rate | intraoperative
whether bad memories exist or not | up to four hours postoperation
  A questionaire about the operation for all parents and children will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, MD, Principal Investigator — Beijing Childrens' Hospital